CLINICAL TRIAL: NCT04230239
Title: A Phase II, Multicentre, Open Label Clinical Trial to Assess the Efficacy and Toxicity of Induction and Consolidation With CPX-351 for Patients Aged 60 to 75 Years With Secondary or High-risk Acute Myeloid Leukemia
Brief Title: Clinical Trial to Assess the Efficacy and Toxicity of Induction and Consolidation With CPX-351 for Patients Aged 60 to 75 Years With Secondary or High-risk Acute Myeloid Leukemia
Acronym: LAMVYX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LAMVYX; 2018-004353-24 (EudraCT Number)
Record Dates: First submitted 2019-11-21; First posted 2020-01-18 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Newly Diagnosed Secondary or High Risk AML
Keywords: Secondary AML; High risk AML
MeSH Terms: interventions — CPX-351

STUDY DESIGN:
Intervention Model Description: This protocol corresponds to a prospective, multicenter, open-label, phase II study to assess efficacy of CPX-351 in elderly patients (60 to 75 years of age) with newly diagnosed high risk AML. In the context of this protocol, a treatment cycle is defined as the first day of study drug administration (Day 1) up to and including the day before the first day of the treatment cycle immediately afterwards. The treatment cycles will begin after Day 42 but no later than Day 80, counting from Day 1 of the treatment cycle immediately before.
  Treatment cycles may be administered while the patient is hospitalized. Patients will receive a maximum of 4 treatment cycles (up to 2 inductions and 2 consolidations) and 6 maintenance cycles. Clinical conditions in the care of patients with acute leukemia require the need for flexibility. However, deviations from the study treatment defined in this section must be prospectively discussed with the coordinator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CPX-351 (Experimental)
  Interventions: Drug: CPX-351

INTERVENTIONS:
Drug: CPX-351 — CPX-351 has IV administration Vyxeos contains 2.2 mg/mL and 5 mg/mL powder for concentrate for solution for infusion of Daunorubicin and cytarabine.
  Each vial contains 44 mg of daunorubicin and 100 mg of cytarabine. After reconstitution, the solution contains 2.2 mg/mL daunorubicin and 5 mg/mL cytarabine

SUMMARY:
This protocol corresponds to a prospective, multicentre, open label, phase II study designed to evaluate the efficacy of CPX-351 in elderly patients with secondary or high-risk AML. The clinical trial is divided into pre-treatment, treatment (induction and consolidation cycles) and follow-up periods and consists of a single arm group. Patients will be enrolled at diagnosis to follow the treatment arm. After that will start induction chemotherapy with CPX-351 regimen (14 days maximum screening period). Once a patient have been evaluated for response and recovered from major complications, he/she will start second course (consolidation 1), unless the bone marrow and peripheral blood assessment is showing less than a complete response, then a second induction may be offered. If a CR or CRi is obtained after the second induction course, patients will start the third course after a rest and recovery period. Patients aged between 60 and 65 years old are recommended to undergo an allo-SCT after first consolidation if they are considered fit for this procedure and they have a full matched related or unrelated donor. Patients aged between 65 and 70 years old can be proposed for an allo-SCT in CR/CRi if they have a composite HSCT co-morbidity index /age less than 4 and a suitable fully matched related donor. In patients over 70 years old, an allo-SCT in first CR should be avoided although the decision should be taken on an individual basis. Patients with CR/CRi who are not considered for an allo-SCT, will follow 6 maintenance cycles with modified courses of CPX-351 schedule. Patients showing unacceptable toxicity along all therapeutic phases that, in consideration of the investigator, will be prematurely discontinued. All patients will be followed-up for survival. The study will be analyzed on an intention to treat basis. Bone marrow and response assessments will be done after each induction and consolidation course, and every 3 months during the first 12 months after starting maintenance therapy. Patients will be followed-up for a minimum period of 1 year after the enrolment of the last patient. Additionally, after the end of the trial, patients will be followed-up for 2 years in order to verify survival and the evolution of the disease. Study design allows a maximum of 59 patients.

DETAILED DESCRIPTION:
This is a prospective, multicenter, open-label, phase II study to assess efficacy of CPX-351 in elderly patients (60 to 75 years of age) with newly diagnosed high risk AML. The study includes a single arm group. The primary endpoint of the study is to assess the CR/CRi rate after induction with CPX-351.

Patients will be enrolled at diagnosis to follow the treatment arm. After that they will start induction chemotherapy with CPX-351 regimen (14 days maximum screening period). Once a patient has been evaluated for response and recovered from major complications (minimum 42 days and maximum 80 days after starting the first course), he/she will start second course (consolidation 1), unless the bone marrow and peripheral blood assessment is showing less than a partial response. If a CR or CRi is obtained after the second course, patients will start the third course after a rest and recovery period (minimum 42 days and maximum 80 days after starting the second course). After the third course an assessment of response will be done.

Patients aged between 60 and 65 years old are recommended to undergo an allo-SCT after first consolidation if they are considered fit for this procedure and they have a full matched related or unrelated donor. Patients with age less than 65-70 years old can be proposed for an allogeneic HSCT in CR/CRi if they have a composite HSCT co-morbidity index /age less than 4 and a suitable fully matched related donor. In patients over 70 years old, an allo-SCT in first CR should be avoided although the decision should be taken on an individual basis.

Patients with CR/CRi who are not considered for an allo-SCT, will follow 6 maintenance cycles with modified courses of CPX-351 schedule. Patients showing unacceptable toxicity along all therapeutic phases that, in consideration of the investigator, will be prematurely discontinued. All patients will be followed-up for survival. The study will be analyzed on an intention to treat basis. Bone marrow and response assessments will be done after each induction and consolidation course, and every 3 months after starting maintenance therapy. Patients will be followed-up for a minimum period of 3 years after the enrollment of the last patient in order to know OS, disease-free, and relapse free survival (RFS), as well as on the duration of remission and cumulative incidence of relapse. Patients may be admitted in hospital to receive the experimental treatment.

The clinical trial is divided into pre-treatment (screening), treatment periods (induction, consolidation and maintenance cycles) and follow-up:

Induction cycle (1 cycle):

It will consist of priming with daily administration of G-CSF on days -1, 1 and 2 (300 mcg/m2/day) subcutaneously, CPX-351 day 1, 3 and 5 (100 units/m2/day) IV in 90 minutes infusion, and subcutaneous G-CSF from day 10 to recovery (5 mg/kg/day). The chemotherapy course may be administered in hospital. If a complete response is obtained after the first cycle of treatment, the patient will receive consolidation cycle. If a partial response is obtained after the first cycle of treatment, the patient will receive induction 2. Response to treatment will be determined by the local investigator and will be the basis for treatment decisions. However, if there is any doubt, it should be discussed with the Study coordinator.

Induction 2 (1 cycle, only for patients with PR after induction 1):

It will consist of priming with daily administration of G-CSF on days -1, 1 and 2 (300 mcg/m2/day) subcutaneously, CPX-351 day 1 and 3 (100 units/m2/day) IV in 90 minutes infusion, and subcutaneous G-CSF from day 10 to recovery (5 mg/kg/day). The chemotherapy course may be administered in hospital.

Consolidation cycle (up to 2 cycles):

It will consist of priming with daily administration of G-CSF on days -1, 1 and 2 (300 mcg/m2/day) subcutaneously, CPX-351 day 1 and 3 (65 units/m2/day) IV in 90 minutes infusion, and subcutaneous G-CSF from day 10 to recovery (5 mg/kg/day). The chemotherapy course may be administered in hospital. Patients aged between 60 and 65 years old are recommended to undergo an allo-SCT after first consolidation if they are considered fit for this procedure and they have a full matched related or unrelated donor. Patients with age between 65-70 years old can be proposed for an allogeneic HSCT in CR/CRi if they have a composite HSCT co-morbidity index /age less than 4 and a suitable fully matched related donor. In patients over 70 years old, an allo-SCT in first CR should be avoided although the decision should be taken on an individual basis.

Maintenance cycle (up to 6 cycles):

For patients in CR and when an allo-SCT is not feasible or recommended, a maintenance treatment could be started for up to 6 additional cycles, on every 4 to 8 weeks courses, according to hematologic recovery.

It will consist of CPX-351 day 1 (50 units/m2/day) IV in 90 minutes infusion. Subcutaneous G-CSF may be used to recovery (5 mg/kg/day) in patients with grade 4 neutropenia and confirmed CR.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent in accordance with national, local, and institutional guidelines. The patient must provide informed consent prior to the first screening procedure. Informed consent form must be signed by the patient and the investigator.
2. Age 60 to 75 years at the time of diagnosis of AML.
3. Newly confirmed diagnosed of AML according to WHO 2008 criteria.
4. Secondary or high risk AML, defined as one of the following:

   * t-AML: documentation of prior cytotoxic therapy or radiation therapy for an unrelated disease in a discharge summary or pharmacy records or radiation therapy records
   * MDSAML: bone marrow documentation of MDS prior to diagnosis of AML (could have been treated previously with hypomethylating or standard chemotherapy)
   * CMMoLAML: bone marrow documentation of CMMoL prior to diagnosis of AML (could have been treated previously with hypomethylating or standard chemotherapy)
   * de novoAML with FISH or cytogenetic changes linked to MDS per WHO 2016 criteria.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
6. Ability to adhere to the study visit schedule and other protocol requirements.
7. Laboratory values fulfilling the following:

   * Serum creatinine < 2.0 mg/mL
   * Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) or total bilirubin < 3 times the upper limit of normal (ULN, subjects with elevated liver enzymes related to disease were instructed to contact the Sponsor) (subjects with Gilbert's Syndrome were instructed to contact the sponsor).
8. Subjects with second malignancies in remission may have been eligible if there was clinical evidence of disease stability for a period ≥ 6 months off cytotoxic chemotherapy, documented by imaging, tumor marker studies at screening. Subjects maintained on long-term nonchemotherapy treatment such as hormonal therapy were eligible.
9. Cardiac ejection fraction ≥ 50% assessed by echocardiography or MUGA.
10. Eligible to receive intensive chemotherapy.
11. Female patients of child-bearing potential must have a negative serum pregnancy test at screening and agree to use reliable methods of contraception for three months after their last dose of medication. Male patients must use a reliable method of contraception (if sexually active with a female of child-bearing potential).
12. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other study procedures

Exclusion Criteria:

1. Patients with genetic diagnosis of acute promyelocytic leukemia.
2. Age <60 years or >75 years.
3. Blastic phase of bcr/abl chronic myeloid leukemia.
4. Patients with de novo AML without FISH or cytogenetic changes linked to MDS per WHO 2016 criteria.
5. Clinical evidence of active central nervous system (CNS) leukemia.
6. Subjects with active (uncontrolled, metastatic) second malignancies.
7. Any major surgery or radiation therapy in 4 weeks.
8. Subjects with myocardial impairment of any cause (eg, cardiomyopathy, ischemic heart disease, significant valvular dysfunction, hypertensive heart disease, and congestive heart failure) resulting in heart failure by New York Heart Association Criteria (Class III or IV staging).
9. Uncontrolled infection; subjects with an infection receiving treatment (antibiotic, antifungal, or antiviral treatment) could be entered into the study provided the subject was respiratory and hemodynamically stable for ≥ 72 hours.
10. Current evidence of invasive fungal infection (blood or tissue culture); subjects with recent fungal infection must have had subsequent negative cultures to be eligible; known HIV (new testing not required) or evidence of active hepatitis B or C infection (with rising transaminase values).
11. Hypersensitivity to cytarabine, daunorubicin or liposomal products.
12. Presence of any severe psychiatric disease or physical condition that, according to the physician´s criteria, contraindicates the inclusion of the patient into the clinical trial.
13. Serum creatinine ≥ 20 mg/dL (unless it is attributable to AML activity).
14. Bilirubin, alkaline phosphatase, or SGOT > 3 times the ULN (unless it is attributable to AML activity).
15. Subjects with prior cumulative anthracycline exposure of greater than 368 mg/m2 daunorubicin (or equivalent).
16. History of Wilson's disease or other copper-metabolism disorder.
17. Patients who have received an investigational agent (for any indication) within 5 half-lives of the agent and until toxicity from this has resolved to grade 1 or less; if the half-life of the agent is unknown, patients must wait 4 weeks prior to first dose of study treatment.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2019-12-26 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-08-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the CR/CRi rate after induction with CPX-351 | After 1 or 2 cycles of induction (between 12 and 16 weeks approximately)
  The primary endpoint of the study is to evaluate the CR/CRi rate after induction with CPX-351. The responses for CR, CRi, PR, therapeutic failure, and disease recurrence are defined for this study based on the revised recommendations of the International Working Group for response criteria.

SECONDARY OUTCOMES:
Incidence of Treatment-Adverse Events (Safety and Tolerability) of the CPX-351 induction regimen. | The induction cycles (up to 2 cycles) will have a mean estimated duration of 6 weeks per cycle. Safety/toxicity assessments will be done in day 1, 8, 15, 22, 29 and 36 of the induction cycles.
  Incidence and description of adverse events occurred during induction regimen.
To evaluate the effect of priming with G-CSF with the CPX-351 regimen | Priming with G-CSF will be done in the induction cycles (up to 2 cycles) and in the consolidation cycles (up to 2 cycles) that will have an an estimated duration of 6 weeks per cycle.
  Differences of leukocytes values (x10^9/L) from baseline values, will be checked in order to know the effect of priming with G-CSF
Incidence of Treatment-Adverse Events (Safety and Tolerability) of the CPX-351 consolidation regimen | Safety/toxicity assessments will be done in day 1, 8, 15, 22, 29 and 36 of the consolidation cycles
  Incidence and description of adverse events occurred during consolidation regimen.
Incidence of Treatment-Adverse Events (Safety and Tolerability) of the CPX-351 maintenance regimen | Safety/toxicity assessments will be done every 2 weeks during the manteinance cycles (24 to 40 weeks of maintenance).
  Incidence and description of adverse events occurred during maintenance regimen.
Overall survival | Estimated 1, 2 and 3 year OS
Event-free, disease-free, and relapse free survival (RFS), as well as on the duration of remission and cumulative incidence of relapse | 1, 2 and 3 years
Incidence of hematologic and non-hematologic adverse events occurred during the study. | At 9 months, which is approximately the estimated mean treatment time.
  Incidence and description of hematologic and non-hematologic adverse events occurred during the study.
To evaluate the impact on the quality of life, using the European Quality of Life-5 Dimensions (EQ5D) form, in patients treated with CPX-351 | The cycles will have a mean estimated duration of 6 weeks and Quality of life questionnaire following EQ-5D will be performed at screening, after induction (day 36), after consolidation 2 ( day 36 of cycle 3) and/or prior to allo-SCT
  European Quality of Life-5 Dimensions (EQ-5D)
To evaluate the impact on the use of medical resources during induction and consolidation phase. | The cycles will have a mean estimated duration of 6 weeks and patients may have up to 2 cycles of induction and up to 2 cycles of consolidation.
  Frequencies and descriptions of medical resources (antibiotics, transfusions, etc)
To evaluate the quality of CR (by study of minimal residual disease percentages in the bone marrow using multiparametric flow cytometry) | After first cycle of induction (6 weeks) and after consolidation 1 (cycle 2: 6 weeks after consolidation 1 onset) only in patients achieving CR/CRi after consolidation 1
To evaluate early mortality (first 60 days) in patients initially treated with CPX-351 | Day 60
To compare the results with a matched-paired historical cohort of the PETHEMA registry | Once the study is completed ( an average of 30 months through study completion)
  Comparison of the different results between patients included in the CPX-351 trial and a retrospective cohort of patients with similarities characteristics at diagnosis (paired analysis). For this purposes, data will be obtained from the retrospective control cohort of the PETHEMA Epidemiologic Registry of Adult AML. Patients will be matched by age (≤65 vs >65, secondary AML vs therapy-related AML vs high-risk according to 2017ELN).
To assess the rate of allo-SCT | After consolidation 1 (aprox 12 weeks) or after consolidation 2 (aprox 18 weeks)
To evaluate 100 day mortality after allo-SCT | 100 day after allo-SCT
To assess compliance of the maintenance schedule | After maintenance (aprox 36 weeks)
  Measure the number and percentage of patients that start maintenance cycles, and how many discontinues during the manteinance phase or complete all manteinance according to protocol

CONTACTS AND LOCATIONS:
Overall Officials: Pau Montesinos Fernández, PhD, Principal Investigator — Hospital Universitario La Fe; José Antonio Pérez Simón, PhD, Principal Investigator — Hospitales Universitarios Virgen del Rocío; Carmen López-Carrero García, Study Chair — Fundación Pethema
Locations (12):
- Spain (12):
  - Institut Català D'Oncologia-Hospital Germans Trias I Pujol, Badalona
  - Institut Català D'Oncologia - Hospital Duran I Reynals, Bellvitge
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario de Gran Canaria Dr. Negrín, Las Palmas
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Ramón Y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital General Del H.U. Virgen Del Rocío, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitario Y Politécnico La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Appelbaum FR, Gundacker H, Head DR, Slovak ML, Willman CL, Godwin JE, Anderson JE, Petersdorf SH. Age and acute myeloid leukemia. Blood. 2006 May 1;107(9):3481-5. doi: 10.1182/blood-2005-09-3724. Epub 2006 Feb 2. PMID 16455952
- [Background] Juliusson G, Antunovic P, Derolf A, Lehmann S, Mollgard L, Stockelberg D, Tidefelt U, Wahlin A, Hoglund M. Age and acute myeloid leukemia: real world data on decision to treat and outcomes from the Swedish Acute Leukemia Registry. Blood. 2009 Apr 30;113(18):4179-87. doi: 10.1182/blood-2008-07-172007. Epub 2008 Nov 13. PMID 19008455
- [Background] Dombret H, Seymour JF, Butrym A, Wierzbowska A, Selleslag D, Jang JH, Kumar R, Cavenagh J, Schuh AC, Candoni A, Recher C, Sandhu I, Bernal del Castillo T, Al-Ali HK, Martinelli G, Falantes J, Noppeney R, Stone RM, Minden MD, McIntyre H, Songer S, Lucy LM, Beach CL, Dohner H. International phase 3 study of azacitidine vs conventional care regimens in older patients with newly diagnosed AML with >30% blasts. Blood. 2015 Jul 16;126(3):291-9. doi: 10.1182/blood-2015-01-621664. Epub 2015 May 18. PMID 25987659
- [Background] Kantarjian HM, Thomas XG, Dmoszynska A, Wierzbowska A, Mazur G, Mayer J, Gau JP, Chou WC, Buckstein R, Cermak J, Kuo CY, Oriol A, Ravandi F, Faderl S, Delaunay J, Lysak D, Minden M, Arthur C. Multicenter, randomized, open-label, phase III trial of decitabine versus patient choice, with physician advice, of either supportive care or low-dose cytarabine for the treatment of older patients with newly diagnosed acute myeloid leukemia. J Clin Oncol. 2012 Jul 20;30(21):2670-7. doi: 10.1200/JCO.2011.38.9429. Epub 2012 Jun 11. PMID 22689805
- [Background] Grimwade D, Walker H, Harrison G, Oliver F, Chatters S, Harrison CJ, Wheatley K, Burnett AK, Goldstone AH; Medical Research Council Adult Leukemia Working Party. The predictive value of hierarchical cytogenetic classification in older adults with acute myeloid leukemia (AML): analysis of 1065 patients entered into the United Kingdom Medical Research Council AML11 trial. Blood. 2001 Sep 1;98(5):1312-20. doi: 10.1182/blood.v98.5.1312. PMID 11520776
- [Background] Frohling S, Schlenk RF, Kayser S, Morhardt M, Benner A, Dohner K, Dohner H; German-Austrian AML Study Group. Cytogenetics and age are major determinants of outcome in intensively treated acute myeloid leukemia patients older than 60 years: results from AMLSG trial AML HD98-B. Blood. 2006 Nov 15;108(10):3280-8. doi: 10.1182/blood-2006-04-014324. Epub 2006 Jul 13. PMID 16840728
- [Background] Tardi P, Johnstone S, Harasym N, Xie S, Harasym T, Zisman N, Harvie P, Bermudes D, Mayer L. In vivo maintenance of synergistic cytarabine:daunorubicin ratios greatly enhances therapeutic efficacy. Leuk Res. 2009 Jan;33(1):129-39. doi: 10.1016/j.leukres.2008.06.028. Epub 2008 Aug 3. PMID 18676016
- [Background] Feldman EJ, Lancet JE, Kolitz JE, Ritchie EK, Roboz GJ, List AF, Allen SL, Asatiani E, Mayer LD, Swenson C, Louie AC. First-in-man study of CPX-351: a liposomal carrier containing cytarabine and daunorubicin in a fixed 5:1 molar ratio for the treatment of relapsed and refractory acute myeloid leukemia. J Clin Oncol. 2011 Mar 10;29(8):979-85. doi: 10.1200/JCO.2010.30.5961. Epub 2011 Jan 31. PMID 21282541
- [Background] Lancet JE, Cortes JE, Hogge DE, Tallman MS, Kovacsovics TJ, Damon LE, Komrokji R, Solomon SR, Kolitz JE, Cooper M, Yeager AM, Louie AC, Feldman EJ. Phase 2 trial of CPX-351, a fixed 5:1 molar ratio of cytarabine/daunorubicin, vs cytarabine/daunorubicin in older adults with untreated AML. Blood. 2014 May 22;123(21):3239-46. doi: 10.1182/blood-2013-12-540971. Epub 2014 Mar 31. PMID 24687088
- [Background] Lancet JE, Uy GL, Cortes JE, et al. Final results of a phase III randomized trial of CPX-351 versus 7+3 in older patients with newly diagnosed high risk (secondary) AML. J Clin Oncol 34, 2016 (suppl; abstr 7000).
- [Background] Cheson BD, Bennett JM, Kopecky KJ, Buchner T, Willman CL, Estey EH, Schiffer CA, Doehner H, Tallman MS, Lister TA, Lo-Coco F, Willemze R, Biondi A, Hiddemann W, Larson RA, Lowenberg B, Sanz MA, Head DR, Ohno R, Bloomfield CD; International Working Group for Diagnosis, Standardization of Response Criteria, Treatment Outcomes, and Reporting Standards for Therapeutic Trials in Acute Myeloid Leukemia. Revised recommendations of the International Working Group for Diagnosis, Standardization of Response Criteria, Treatment Outcomes, and Reporting Standards for Therapeutic Trials in Acute Myeloid Leukemia. J Clin Oncol. 2003 Dec 15;21(24):4642-9. doi: 10.1200/JCO.2003.04.036. PMID 14673054
- [Background] Lee SJ, Lindquist K, Segal MR, Covinsky KE. Development and validation of a prognostic index for 4-year mortality in older adults. JAMA. 2006 Feb 15;295(7):801-8. doi: 10.1001/jama.295.7.801. PMID 16478903
- [Background] Dohner H, Estey E, Grimwade D, Amadori S, Appelbaum FR, Buchner T, Dombret H, Ebert BL, Fenaux P, Larson RA, Levine RL, Lo-Coco F, Naoe T, Niederwieser D, Ossenkoppele GJ, Sanz M, Sierra J, Tallman MS, Tien HF, Wei AH, Lowenberg B, Bloomfield CD. Diagnosis and management of AML in adults: 2017 ELN recommendations from an international expert panel. Blood. 2017 Jan 26;129(4):424-447. doi: 10.1182/blood-2016-08-733196. Epub 2016 Nov 28. PMID 27895058
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Derived] Rodriguez-Arboli E, Rodriguez-Veiga R, Soria-Saldise E, Bergua JM, Caballero-Velazquez T, Arnan M, Vives S, Serrano J, Bernal T, Martinez-Sanchez P, Tormo M, Rodriguez-Medina C, Herrera-Puente P, Lavilla-Rubira E, Boluda B, Acuna-Cruz E, Cano I, Caceres S, Ballesteros J, Falantes J, Martinez-Cuadron D, Perez-Simon JA, Montesinos P; PETHEMA Group. A phase 2, multicenter, clinical trial of CPX-351 in older patients with secondary or high-risk acute myeloid leukemia: PETHEMA-LAMVYX. Cancer. 2025 Jan 1;131(1):e35618. doi: 10.1002/cncr.35618. Epub 2024 Oct 30. PMID 39476204